CLINICAL TRIAL: NCT02399527
Title: Lymphatic Anomalies Registry for the Assessment of Outcome Data
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Lymphatic Malformation Institute (Other)
Responsible Party: Principal Investigator, Melisa Ruiz-Gutierrez, Attending Physician - Pediatric Hematology/Oncology, Boston Children's Hospital
Other Study IDs: P00007182
Record Dates: First submitted 2015-03-17; First posted 2015-03-26 (Estimated); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Lymphatic Malformation; Generalized Lymphatic Anomaly (GLA); Central Conducting Lymphatic Anomaly; CLOVES Syndrome; Gorham-Stout Disease ("Disappearing Bone Disease"); Blue Rubber Bleb Nevus Syndrome; Kaposiform Lymphangiomatosis; Kaposiform Hemangioendothelioma/Tufted Angioma; Klippel-Trenaunay Syndrome; Lymphangiomatosis
Keywords: Vascular Anomalies; Lymphatic Anomalies; Lymphatic Malformation
MeSH Terms: conditions — Lymphatic Abnormalities; Congenital Lipomatous Overgrowth, Vascular Malformations, and Epidermal Nevi; Osteolysis, Essential; Blue rubber bleb nevus syndrome; Kaposiform Hemangioendothelioma; Tufted angioma; Klippel-Trenaunay-Weber Syndrome; Vascular Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Lymphatic anomalies are a rare subset of vascular anomalies that are poorly understood. the understanding of the natural history, long-term outcomes, risk factors for morbidity and mortality, and the relative benefit of medical therapies and procedures is limited.The goal of this project is to better understand these diseases and improve the care of theses rare patients. To do this, the investigators are conducting an observational study of patients with lymphatic anomalies, including an annual follow-up questionnaire to gather prospective data on mortality, morbidity, treatments, and functionality as well as quality of life.

DETAILED DESCRIPTION:
The purpose of the Lymphatic Anomalies Registry, created at Boston Children's Hospital, is to create a database to help current and future patients diagnosed with a lymphatic anomaly. The ultimate goal of the registry is to better understand and predict responses to therapies and risk factors for complications. Although the Lymphatic Anomalies Registry exists at Boston Children's Hospital, patients can be entered into the registry regardless of whether or not they visit Boston Children's Hospital, thus increasing the program's accessibility. The Lymphatic Anomalies Registry includes patients who have vascular anomalies with a lymphatic component across various diagnoses. From the patient's perspective, participation in the Lymphatic Anomalies Registry means taking part in a short, thirty minute interview, and providing the registry with access to medical records. The interview is conducted verbally with study staff of the Lymphatic Anomalies Registry, and can take place either at the hospital, or over the phone. During the interview, the registry will inquire about the patient's diagnosis, disease features, medical therapies, and procedures. Interested prospective patients will receive an introductory packet from the registry with information on how to proceed in the registry process. All obtained patient information is housed on a secure, HIPPA compliant, internal database, managed by Boston Children's Hospital staff. Patient information entered into the external database is de-identified. The research teams will also obtain a medical record release form to request the patient's medical record for review in our study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of complex vascular tumor, malformation or overgrowth syndrome with significant lymphatic component

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both domestic and international patients with complex lymphatic anomalies, as described above, are eligible to participate. Travel to Boston is not required for participation. Eligible patients are identified through active referral in the Vascular Anomalies Center at Boston Children's Hospital. Physicians and patients may also refer eligible patients directly to the Lymphatic Anomalies Registry. Patients may indicate interest in participation themselves by contacting the registry team through the "Contact Us" link on www.lymphaticregistry.org.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2035-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
To characterize the heterogeneity of lymphatic disorders, including demographics, presentation, and complications. | 15 years
To identify factors that are prognostic of the occurrence of complications, including effusions, coagulopathy, ectatic draining veins, prior infections, visceral involvement, bone involvement, and development of cardiopulmonary symptoms. | 15 years
To identify factors prognostic of poor outcome and use them to develop "staging" of lymphatic anomalies. | 15 years
To describe the natural history of lymphatic anomalies, including morbidity and mortality. | 15 years
To describe the therapies (medical and procedural), adverse events and responses to therapy in patients with lymphatic anomalies. | 15 years
To pilot quality of life, functional assessment and pain scoring tools in this patient population. | 15 years

SECONDARY OUTCOMES:
To estimate the proportion of time that patients with lymphatic anomalies have affected offspring. | 15 years
To assess for correlations of pregnancy complications or medications taken during pregnancy with the development of lymphatic anomalies. | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Melisa Ruiz-Gutierrez, M.D., Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Rankin H, Zwicker K, Trenor CC 3rd. Caution is recommended prior to sildenafil use in vascular anomalies. Pediatr Blood Cancer. 2015 Nov;62(11):2015-7. doi: 10.1002/pbc.25600. Epub 2015 May 15. PMID 25982365
- [Result] Croteau SE, Kozakewich HP, Perez-Atayde AR, Fishman SJ, Alomari AI, Chaudry G, Mulliken JB, Trenor CC 3rd. Kaposiform lymphangiomatosis: a distinct aggressive lymphatic anomaly. J Pediatr. 2014 Feb;164(2):383-8. doi: 10.1016/j.jpeds.2013.10.013. Epub 2013 Nov 16. PMID 24252784
- [Result] Strychowsky JE, Rahbar R, O'Hare MJ, Irace AL, Padua H, Trenor CC 3rd. Sirolimus as treatment for 19 patients with refractory cervicofacial lymphatic malformation. Laryngoscope. 2018 Jan;128(1):269-276. doi: 10.1002/lary.26780. Epub 2017 Aug 7. PMID 28782106
- See also: Lymphatic Anomalies Registry Study Info — https://www.childrenshospital.org/programs/lymphatic-anomalies-registry